CLINICAL TRIAL: NCT06297187
Title: A Retrospective Registry on the Use of CUSA® for the Treatment of Vulvar Intraepithelial Neoplasia (VIN) and Condyloma Acuminata
Brief Title: Cavitronic Ultrasonic Surgical Aspiration (CUSA) Women's Health Study
Status: Completed | Type: Observational
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: C-CUSAWH-001
Record Dates: First submitted 2024-02-27; First posted 2024-03-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Vulvar Intraepithelial Neoplasia; Condylomata Acuminata
Keywords: Gynecologic Oncology; VIN; Vulvar Intraepithelial Neoplasia; Condylomata Acuminata
MeSH Terms: conditions — Condylomata Acuminata

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- CUSA Excel®: Subjects having had treatment for Vulvar Intraepithelial Neoplasia (VIN) and/or condyloma acuminata using CUSA® Excel system.
  Interventions: Device: CUSA (Cavitronic Ultrasonic Surgical Aspirator)
- CUSA Clarity®: Subject having had treatment for Vulvar Intraepithelial Neoplasia (VIN) and/or condyloma acuminata using CUSA® Clarity system.
  Interventions: Device: CUSA (Cavitronic Ultrasonic Surgical Aspirator)

INTERVENTIONS:
Device: CUSA (Cavitronic Ultrasonic Surgical Aspirator) — CUSA® Excel and CUSA® Clarity Ultrasonic Surgical Aspirator Systems are indicated for use in the surgical procedures where fragmentation, emulsification and aspiration of soft and hard tissue is desirable.

SUMMARY:
The study is a single arm, retrospective, single-center, post market registry.

The purpose of this Registry is to collect data to demonstrate the safety and performance of CUSA® for the treatment of Vulvar Intraepithelial Neoplasia (VIN) and condyloma acuminata.

DETAILED DESCRIPTION:
CUSA® Excel/Clarity Ultrasonic Surgical Aspirator System is indicated for use in the following surgical procedures where fragmentation, emulsification and aspiration of soft and hard tissue is desirable:

* Neurosurgery
* Gastrointestinal and affiliated organ surgery
* Urological surgery
* General surgery
* Orthopedic surgery
* Gynecological surgery
* Laparoscopic surgery

This Registry adds data to support the safety and efficacy for a gynecological surgery indication expansion for the use of CUSA in Vulvar Intraepithelial Neoplasia (VIN) and condyloma acuminata.

Information obtained from this retrospective Registry will help inform a potential future prospective study for this indication in a real-world population.

ELIGIBILITY:
Inclusion Criteria:

* Subject had been diagnosed with primary or recurrent Vulvar Intraepithelial Neoplasia (VIN) or condyloma acuminata, treated with CUSA and confirmed by a CUSA pathology report.
* Subject had post-operative visits completed at the gynecologic oncology practice.
* Subject had surgery with CUSA between January 2010 and December 2022.

Exclusion Criteria: Not Applicable

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients identified as genetically female at birth.
Study Population: Patients identified as genetically female at birth between the ages of 18 and greater (inclusive) at the time they underwent treatment with CUSA for Vulvar Intraepithelial Neoplasia (VIN) or condyloma acuminata between January 2010 and December 2022. Pregnant patients will be included.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2024-02-23 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Proportion of Subjects with Complete Removal of Vulvar Intraepithelial Neoplasia and condyloma acuminata | During Surgery
  Ability of CUSA to completely remove Vulvar Intraepithelial Neoplasia (VIN) and condyloma acuminata.

SECONDARY OUTCOMES:
Primary Site Recurrence | Up to 12 months Postoperatively.
  Incidence of Primary Site Recurrence of Vulvar Intraepithelial Neoplasia or condyloma acuminata.

CONTACTS AND LOCATIONS:
Overall Officials: DeEtte Vasques, DO, Principal Investigator — Private Practice, Dallas, Texas
Locations (1):
- The Center for Cancer and Blood Disorders, Dallas, Texas, United States